CLINICAL TRIAL: NCT04998097
Title: Changes in Serum miRNA and BDNF Levels in Bipolar II Depression Treated by Theta-burst Stimulation: A Randomized Sham-controlled Exploratory Study
Brief Title: The Role of iTBS in Bipolar II Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Sheng Yu Lee, Attending physician, Department of Psychiatry, Kaohsiung Veterans General Hospital, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-CT3-23(210303-1)
Record Dates: First submitted 2021-07-01; First posted 2021-08-10 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Bipolar II Disorder, Most Recent Episode Major Depressive
Keywords: rTMS; BDNF; micro RNA; cognitive function
MeSH Terms: conditions — Bipolar Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: one experimental and one sham group
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (iTBS group) (Experimental): device: Magstim Rapid2 Stimulator
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)
- sham group (Sham Comparator): device shame Magstim Rapid2 Stimulator
  Interventions: Device: sham repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation (rTMS) — Investigators adopted the iTBS protocol which follows the standard TBS protocols, with 3-pulse 50-Hz bursts given every 200 ms (at 5 Hz) and an intensity of 80% motor threshold. In each session, a 2-s train of bursts will be repeated every 10 s for a total of 570 s (1800 pulses) to the left dorsolateral prefrontal cortex (DLPFC). TBS sessions will be scheduled daily in a 5-day sequence, for a total of 10 sessions in 2 weeks.
  Arms: experimental (iTBS group)
Device: sham repetitive transcranial magnetic stimulation (rTMS) — no stimulation, Sham TBS sessions will be scheduled daily in a 5-day sequence, for a total of 10 sessions in 2 weeks.
  Arms: sham group

SUMMARY:
There is a paucity of evidence-supported treatment choices for bipolar II depression (BD-II depression), hindered by multiple comorbidity and manic switch. In addition, a slower response also burdens the patients. Intermittent theta-burst stimulation (iTBS) is a new form of Repetitive transcranial magnetic stimulation (rTMS) which is more powerful and requires less time of operation (i.e., about 1/3 of traditional treatment time) compared to traditional rTMS protocols. The antidepressant effect of iTBS for major depressive disorder is well established; however, its effect for BD-II depression is still undetermined with few investigations. In the current study, the investigators plan to conduct a randomized, controlled study to directly compare antidepressant effects of iTBS (n=30) versus sham (n=30) for BD-II depression under treatment of quetiapine monotherapy. The participants will receive 10 times of iTBS sessions in 2 weeks (daily from Monday to Friday and off on the weekends for 2 weeks), followed on the end of week 2 (right after treatment,), week 6 and week 12. The investigators hypothesize that iTBS is effective for BD-II depression and may improve cognitive decline associated with BD-II. In addition, the investigators have identified several microRNAs (miRNAs) (miR-7-5p, miR-142-3p, miR-221-5p, and miR-370-3p) which may aid the diagnosis of BD-II and such diagnostic model was patented in Taiwan. The investigators further found significant correlations with these miRNAs with peripheral levels of brain derived neurotrophic factor (BDNF). The investigators inferred that these miRNAs may be associated with susceptibility with BD-II thru modulation of BDNF. Because modulation of BDNF level is one of the anti-depression mechanism for rTMS, the investigators plan to monitor the changes of these candidate miRNAs and BDNF levels in serum before and after iTBS treatment (week 0, 2,6,12), in attempt to clarify whether these miRNAs may be treatment biomarker as well. The investigators believe that the current study result may be a great addition for predictor for therapeutic assessment and precision treatment of BD-II depression.

DETAILED DESCRIPTION:
In this 2-year prospective, randomized, and controlled study, the investigators plan to recruit a total of 60 patients with BD-II depression. According to a random distribution table, the participants will be randomly divided into the two subgroups, respectively: the real iTBS group (n=30) and the sham iTBS group (n=30). Patients with BD-II depression between 20 and 65 years old will be recruited in 2 years. Patients will be evaluated by research psychiatrists after a thorough medical and neurological workup. The Chinese Version of Modified Schedule of Affective Disorder and Schizophrenia-Life Time (SADS-L) will be conducted for confirmation of the diagnosis. Although DSM-IV-TR criteria require a minimum duration of 4 days of hypomania, current epidemiologic data suggest that a 2-day duration is more prevalent in community samples; therefore, the investigators will use the 2-day minimum for hypomania in the diagnosis of BD-II. Eligible participants, aged 20-65, need to have a DSM-IV-TR diagnosis of BD-II. HDRS and YMRS will be used to evaluate severity of mood symptoms. Only patients in depressive state (HDRS≧18) will be recruited. Inclusion criteria are those with diagnosis of BD-II either first-onset or with previous episodes. Exclusion criteria are (i) any DSM-IV-TR Axis I diagnosis, including organic mental disorders, substance use disorder, and other major and minor mental illnesses other than BD-II, (ii) any significant medical illness, (iii) any neurological disorders, and (iv) any poorly controlled physical illness that might influence the interview and study results; (v) any form of metal implants; (iv) any history of seizures, or medications known to lower seizure threshold; (vii) history of exposure to rTMS or electroconvulsive therapy.

During the course of the follow-up, all patients will receive open-label quetiapine adjusted individually according to the clinical response and side effects in the first two weeks and will be maintained till the end of the trial, with the final dose ranging from 200 to 700 mg/d. Concomitant benzodiazepine medication (lorazepam < 4 mg) may be used for insomnia during the study. No other antidepressants, mood stabilizers, first or second-generation antipsychotics will be allowed during the study.

Twenty milliliters of whole blood will be withdrawn from the antecubital vein of each participant and prepared as serum for the purpose of total RNA extraction and for level of BDNF analysis.

The patients will be followed for 12 weeks and blood samples (20cc whole blood) and clinical symptoms will be examined at week0, the end of week 2, 6 and week 12.

Clinical severity will be assessed by the HDRS and YMRS and Clinical ratings will be performed by research psychiatrists who are trained and experienced in the rating scales. Assessments will be performed after recruitment, week 0 and on the end of week 2, 6, and 12. RNA extraction Serum will be isolated from the whole blood and stored at -80°C immediately.

The miRNeasy kit (Qiagen, CA) will be implemented for total RNA extraction using serum from all patients and controls.

Total RNAs will be isolated from 250-µL serum of clinical samples and subjected to quantitative detection of miRNA by using the cDNA TaqMan Advanced miRNA cDNA synthesis kit (Applied Biosystems, Inc., USA). Synthesized cDNA samples will then be subjected to qRT-PCR by using the TaqManR Universal PCR Master Mix II and TaqMan Advanced miRNA assays according to manufacturer's instructions (Applied Biosystems). Expression levels of miRNAs in serum will be normalized with miR-16. The following IDs of miRNA will be used: hsa-miR-7-5p (483061_mir), hsa-miR-142-3p (477910_mir), hsa-miR-370-3p (478326_mir), and hsa-miR-221-5p (478778_mir), and has-miR-16 (481312_mir).

The level of plasma BDNF will be measured by a BDNF kit (Quantikine Human BDNF kit; R&D Systems, Minneapolis, MN) and an enzyme-linked immunosorbent assay (ELISA) reader (SpectraMax-M2; Molecular Devices, Sunnyvale, CA) which has a minimum detectable dose of 80 pg/ml.

All iTBS procedures will be conducted in the Department of Psychiatry in Kaohsiung Veterans General Hospital. An Magstim Rapid2 stimulator with eight-figure coil was used for stimulation. The resting motor threshold (MT) will be determined by the minimum intensity of magnetic stimulation on the primary motor cortex to elicit five visible muscle contractions out of ten consecutive stimuli in the contralateral abductor pollicis brevis muscle . Because a recent meta-analysis found that low stimulation intensities, high number of pulses per session, short treatment periods (less or equal to 2 weeks), and intermittent TBS (iTBS) might be the optimal parameters of TBS protocols, investigators adopted the iTBS protocol which follows the standard TBS protocols, with 3-pulse 50-Hz bursts given every 200 ms (at 5 Hz) and an intensity of 80% motor threshold. In each session, a 2-s train of bursts will be repeated every 10 s for a total of 570 s (1800 pulses) to the left dorsolateral prefrontal cortex (DLPFC). TBS sessions will be scheduled daily in a 5-day sequence, for a total of 10 sessions in 2 weeks. The figure-eight coil will be positioned in a para-sagittal plane 5.5 cm anterior to the site of MT determination and magnetic stimulation will be consequently delivered to the brain region of left DLPFC. Finally, after the 2-week double-blind phase of active or sham iTBS treatment, each patient will be followed at week 6 and week 12 to evaluate the response to the iTBS treatment.

Neuropsychological function assessment Brief Assessment of Cognition in Affective Disorders (BACA) Investigators will adopt the BACA to evaluate objective cognitive functioning in patients with mood disorders. This instrument consists of seven subtests, including Verbal Memory (List Learning), Working Memory (Digit Sequencing), Processing Speed (Verbal Fluency; Token Motor Task; Symbol Coding), Reasoning and Problem Solving (Tower of London [TOL]), and tests of affective interference (emotional distractibility and affective memory) and emotional disinhibition, which are then summed up as affective composite scores. This assessment takes approximately 45 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. The Chinese Version of Modified Schedule of Affective Disorder and Schizophrenia-Life Time (SADS-L) and DSM-IV-TR will be conducted for confirmation of the diagnosis of BD-II.
2. Aged 20-65.
3. HDRS and YMRS will be used to evaluate severity of mood symptoms. Only patients in deressive state (HDRS≧18) will be recruited.

Exclusion Criteria:

1. Any DSM-IV-TR Axis I diagnosis, including organic mental disorders, substance use disorder, and other major and minor mental illnesses other than BD-II.
2. Any significant medical illness.
3. Any neurological disorders.
4. Any poorly controlled physical illness that might influence the interview and study results.
5. Any form of metal implants.
6. Any history of seizures, or medications known to lower seizure threshold.
7. History of exposure to TMS or electroconvulsive therapy.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS) | Baseline, week 2 (after rTMS intervention), week6, week 12 (endpoint).
  Clinical depression severity will be assessed by the HDRS. The total score range is from 0 to 52. Higher scores (>=18) indicate a greater degree of depression. A significant change in the score is considered a response to rTMS. HDRS will be assessed from baseline, week2, week 6,and week12.

SECONDARY OUTCOMES:
Young Mania Rating Scale (YMRS) | Baseline, week 2 (after rTMS intervention), week6, week 12 (endpoint).
  Clinical manic severity will be assessed by the YMRS. The total score range is from 0 to 44. Higher scores (>29) indicate a greater degree of maina. YMRS will be used to assess mood severity at baseline, week2, week6,and week12..

OTHER OUTCOMES:
Brief Assessment of Cognition in Affective Disorders (BACA) | Baseline, endpoint (week 12)
  The BACA is used to evaluate objective cognitive functioning in patients with mood disorders. A T-score of 50 demonstrates average functioning with regard to the healthy population with the same age and gender; the standard deviation is 10 points.
plasma miRNA | Baseline, week 2 (after rTMS intervention), week6, week 12 (endpoint).
  The following plasma miRNA levels: miR-7-5-p, miR-142-3p, miR-370-3p, miR221-5p (miRNA unit: delta Ct).
plasma BDNF level | Baseline, week 2 (after rTMS intervention), week6, week 12 (endpoint).
  Plasma BDNF levels.

CONTACTS AND LOCATIONS:
Locations (1):
- KaohsiungVGH, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Angst J, Gamma A, Benazzi F, Ajdacic V, Eich D, Rossler W. Toward a re-definition of subthreshold bipolarity: epidemiology and proposed criteria for bipolar-II, minor bipolar disorders and hypomania. J Affect Disord. 2003 Jan;73(1-2):133-46. doi: 10.1016/s0165-0327(02)00322-1. PMID 12507746
- [Background] Benazzi F, Akiskal HS. Refining the evaluation of bipolar II: beyond the strict SCID-CV guidelines for hypomania. J Affect Disord. 2003 Jan;73(1-2):33-8. doi: 10.1016/s0165-0327(02)00327-0. PMID 12507735
- [Background] Akiskal HS, Pinto O. The evolving bipolar spectrum. Prototypes I, II, III, and IV. Psychiatr Clin North Am. 1999 Sep;22(3):517-34, vii. doi: 10.1016/s0193-953x(05)70093-9. PMID 10550853
- [Background] Phillips ML, Kupfer DJ. Bipolar disorder diagnosis: challenges and future directions. Lancet. 2013 May 11;381(9878):1663-71. doi: 10.1016/S0140-6736(13)60989-7. PMID 23663952
- [Background] Vieta E, Berk M, Schulze TG, Carvalho AF, Suppes T, Calabrese JR, Gao K, Miskowiak KW, Grande I. Bipolar disorders. Nat Rev Dis Primers. 2018 Mar 8;4:18008. doi: 10.1038/nrdp.2018.8. PMID 29516993
- [Background] Carvalho AF, Firth J, Vieta E. Bipolar Disorder. N Engl J Med. 2020 Jul 2;383(1):58-66. doi: 10.1056/NEJMra1906193. No abstract available. PMID 32609982
- [Background] Judd LL, Akiskal HS. Depressive episodes and symptoms dominate the longitudinal course of bipolar disorder. Curr Psychiatry Rep. 2003 Dec;5(6):417-8. doi: 10.1007/s11920-003-0077-2. No abstract available. PMID 14609495
- [Background] Mosolov S, Ushkalova A, Kostukova E, Shafarenko A, Alfimov P, Kostyukova A, Angst J. Bipolar II disorder in patients with a current diagnosis of recurrent depression. Bipolar Disord. 2014 Jun;16(4):389-99. doi: 10.1111/bdi.12192. Epub 2014 Mar 1. PMID 24580856
- [Background] Earley W, Burgess MV, Rekeda L, Dickinson R, Szatmari B, Nemeth G, McIntyre RS, Sachs GS, Yatham LN. Cariprazine Treatment of Bipolar Depression: A Randomized Double-Blind Placebo-Controlled Phase 3 Study. Am J Psychiatry. 2019 Jun 1;176(6):439-448. doi: 10.1176/appi.ajp.2018.18070824. Epub 2019 Mar 8. PMID 30845817
- [Background] Nierenberg AA, McIntyre RS, Sachs GS. Improving outcomes in patients with bipolar depression: a comprehensive review. J Clin Psychiatry. 2015 Mar;76(3):e10. doi: 10.4088/JCP.13091ip1. PMID 25830453
- [Background] El-Mallakh RS, Vohringer PA, Ostacher MM, Baldassano CF, Holtzman NS, Whitham EA, Thommi SB, Goodwin FK, Ghaemi SN. Antidepressants worsen rapid-cycling course in bipolar depression: A STEP-BD randomized clinical trial. J Affect Disord. 2015 Sep 15;184:318-21. doi: 10.1016/j.jad.2015.04.054. Epub 2015 Jun 10. PMID 26142612
- [Background] Rossini PM, Rossi S. Transcranial magnetic stimulation: diagnostic, therapeutic, and research potential. Neurology. 2007 Feb 13;68(7):484-8. doi: 10.1212/01.wnl.0000250268.13789.b2. PMID 17296913
- [Background] Hett D, Marwaha S. Repetitive Transcranial Magnetic Stimulation in the Treatment of Bipolar Disorder. Ther Adv Psychopharmacol. 2020 Nov 18;10:2045125320973790. doi: 10.1177/2045125320973790. eCollection 2020. PMID 33282175
- [Background] Goldwaser EL, Daddario K, Aaronson ST. A retrospective analysis of bipolar depression treated with transcranial magnetic stimulation. Brain Behav. 2020 Dec;10(12):e01805. doi: 10.1002/brb3.1805. Epub 2020 Nov 10. PMID 33169946
- [Background] McGirr A, Karmani S, Arsappa R, Berlim MT, Thirthalli J, Muralidharan K, Yatham LN. Clinical efficacy and safety of repetitive transcranial magnetic stimulation in acute bipolar depression. World Psychiatry. 2016 Feb;15(1):85-6. doi: 10.1002/wps.20300. No abstract available. PMID 26833619
- [Background] Daskalakis ZJ. Theta-burst transcranial magnetic stimulation in depression: when less may be more. Brain. 2014 Jul;137(Pt 7):1860-2. doi: 10.1093/brain/awu123. Epub 2014 May 15. No abstract available. PMID 24833712
- [Background] Blumberger DM, Vila-Rodriguez F, Thorpe KE, Feffer K, Noda Y, Giacobbe P, Knyahnytska Y, Kennedy SH, Lam RW, Daskalakis ZJ, Downar J. Effectiveness of theta burst versus high-frequency repetitive transcranial magnetic stimulation in patients with depression (THREE-D): a randomised non-inferiority trial. Lancet. 2018 Apr 28;391(10131):1683-1692. doi: 10.1016/S0140-6736(18)30295-2. Epub 2018 Apr 26. PMID 29726344
- [Background] Li CT, Cheng CM, Chen MH, Juan CH, Tu PC, Bai YM, Jeng JS, Lin WC, Tsai SJ, Su TP. Antidepressant Efficacy of Prolonged Intermittent Theta Burst Stimulation Monotherapy for Recurrent Depression and Comparison of Methods for Coil Positioning: A Randomized, Double-Blind, Sham-Controlled Study. Biol Psychiatry. 2020 Mar 1;87(5):443-450. doi: 10.1016/j.biopsych.2019.07.031. Epub 2019 Aug 9. PMID 31563272
- [Background] Li CT, Chen MH, Juan CH, Huang HH, Chen LF, Hsieh JC, Tu PC, Bai YM, Tsai SJ, Lee YC, Su TP. Efficacy of prefrontal theta-burst stimulation in refractory depression: a randomized sham-controlled study. Brain. 2014 Jul;137(Pt 7):2088-98. doi: 10.1093/brain/awu109. Epub 2014 May 10. PMID 24817188
- [Background] Luan D, Zhao MG, Shi YC, Li L, Cao YJ, Feng HX, Zhang ZJ. Mechanisms of repetitive transcranial magnetic stimulation for anti-depression: Evidence from preclinical studies. World J Psychiatry. 2020 Oct 19;10(10):223-233. doi: 10.5498/wjp.v10.i10.223. eCollection 2020 Oct 19. PMID 33134113
- [Background] Chen YH, Zhang RG, Xue F, Wang HN, Chen YC, Hu GT, Peng Y, Peng ZW, Tan QR. Quetiapine and repetitive transcranial magnetic stimulation ameliorate depression-like behaviors and up-regulate the proliferation of hippocampal-derived neural stem cells in a rat model of depression: The involvement of the BDNF/ERK signal pathway. Pharmacol Biochem Behav. 2015 Sep;136:39-46. doi: 10.1016/j.pbb.2015.07.005. Epub 2015 Jul 12. PMID 26176197
- [Background] Pasquinelli AE. MicroRNAs and their targets: recognition, regulation and an emerging reciprocal relationship. Nat Rev Genet. 2012 Mar 13;13(4):271-82. doi: 10.1038/nrg3162. PMID 22411466
- [Background] Saba R, Schratt GM. MicroRNAs in neuronal development, function and dysfunction. Brain Res. 2010 Jun 18;1338:3-13. doi: 10.1016/j.brainres.2010.03.107. Epub 2010 Apr 7. PMID 20380818
- [Background] Magill ST, Cambronne XA, Luikart BW, Lioy DT, Leighton BH, Westbrook GL, Mandel G, Goodman RH. microRNA-132 regulates dendritic growth and arborization of newborn neurons in the adult hippocampus. Proc Natl Acad Sci U S A. 2010 Nov 23;107(47):20382-7. doi: 10.1073/pnas.1015691107. Epub 2010 Nov 8. PMID 21059906
- [Background] Moreau MP, Bruse SE, David-Rus R, Buyske S, Brzustowicz LM. Altered microRNA expression profiles in postmortem brain samples from individuals with schizophrenia and bipolar disorder. Biol Psychiatry. 2011 Jan 15;69(2):188-93. doi: 10.1016/j.biopsych.2010.09.039. PMID 21183010
- [Background] Wang Z, Zhang C, Huang J, Yuan C, Hong W, Chen J, Yu S, Xu L, Gao K, Fang Y. MiRNA-206 and BDNF genes interacted in bipolar I disorder. J Affect Disord. 2014 Jun;162:116-9. doi: 10.1016/j.jad.2014.03.047. Epub 2014 Apr 3. PMID 24767015
- [Background] Ha TY. The Role of MicroRNAs in Regulatory T Cells and in the Immune Response. Immune Netw. 2011 Feb;11(1):11-41. doi: 10.4110/in.2011.11.1.11. Epub 2011 Feb 28. PMID 21494372
- [Background] Bocchio-Chiavetto L, Maffioletti E, Bettinsoli P, Giovannini C, Bignotti S, Tardito D, Corrada D, Milanesi L, Gennarelli M. Blood microRNA changes in depressed patients during antidepressant treatment. Eur Neuropsychopharmacol. 2013 Jul;23(7):602-11. doi: 10.1016/j.euroneuro.2012.06.013. Epub 2012 Aug 25. PMID 22925464
- [Background] Lee SY, Lu RB, Wang LJ, Chang CH, Lu T, Wang TY, Tsai KW. Serum miRNA as a possible biomarker in the diagnosis of bipolar II disorder. Sci Rep. 2020 Jan 24;10(1):1131. doi: 10.1038/s41598-020-58195-0. PMID 31980721
- [Background] Soeiro-de-Souza MG, Dias VV, Figueira ML, Forlenza OV, Gattaz WF, Zarate CA Jr, Machado-Vieira R. Translating neurotrophic and cellular plasticity: from pathophysiology to improved therapeutics for bipolar disorder. Acta Psychiatr Scand. 2012 Nov;126(5):332-41. doi: 10.1111/j.1600-0447.2012.01889.x. Epub 2012 Jun 8. PMID 22676371
- [Background] Lim CS, Baldessarini RJ, Vieta E, Yucel M, Bora E, Sim K. Longitudinal neuroimaging and neuropsychological changes in bipolar disorder patients: review of the evidence. Neurosci Biobehav Rev. 2013 Mar;37(3):418-35. doi: 10.1016/j.neubiorev.2013.01.003. Epub 2013 Jan 12. PMID 23318228
- [Background] Monteggia LM, Barrot M, Powell CM, Berton O, Galanis V, Gemelli T, Meuth S, Nagy A, Greene RW, Nestler EJ. Essential role of brain-derived neurotrophic factor in adult hippocampal function. Proc Natl Acad Sci U S A. 2004 Jul 20;101(29):10827-32. doi: 10.1073/pnas.0402141101. Epub 2004 Jul 12. PMID 15249684
- [Background] Cotman CW, Berchtold NC. Exercise: a behavioral intervention to enhance brain health and plasticity. Trends Neurosci. 2002 Jun;25(6):295-301. doi: 10.1016/s0166-2236(02)02143-4. PMID 12086747
- [Background] Hofer M, Pagliusi SR, Hohn A, Leibrock J, Barde YA. Regional distribution of brain-derived neurotrophic factor mRNA in the adult mouse brain. EMBO J. 1990 Aug;9(8):2459-64. doi: 10.1002/j.1460-2075.1990.tb07423.x. PMID 2369898
- [Background] de Oliveira GS, Cereser KM, Fernandes BS, Kauer-Sant'Anna M, Fries GR, Stertz L, Aguiar B, Pfaffenseller B, Kapczinski F. Decreased brain-derived neurotrophic factor in medicated and drug-free bipolar patients. J Psychiatr Res. 2009 Sep;43(14):1171-4. doi: 10.1016/j.jpsychires.2009.04.002. Epub 2009 May 26. PMID 19473667
- [Background] Fernandes BS, Gama CS, Cereser KM, Yatham LN, Fries GR, Colpo G, de Lucena D, Kunz M, Gomes FA, Kapczinski F. Brain-derived neurotrophic factor as a state-marker of mood episodes in bipolar disorders: a systematic review and meta-regression analysis. J Psychiatr Res. 2011 Aug;45(8):995-1004. doi: 10.1016/j.jpsychires.2011.03.002. Epub 2011 May 6. PMID 21550050
- [Background] Molendijk ML, Spinhoven P, Polak M, Bus BA, Penninx BW, Elzinga BM. Serum BDNF concentrations as peripheral manifestations of depression: evidence from a systematic review and meta-analyses on 179 associations (N=9484). Mol Psychiatry. 2014 Jul;19(7):791-800. doi: 10.1038/mp.2013.105. Epub 2013 Aug 20. PMID 23958957
- [Background] Kauer-Sant'Anna M, Kapczinski F, Andreazza AC, Bond DJ, Lam RW, Young LT, Yatham LN. Brain-derived neurotrophic factor and inflammatory markers in patients with early- vs. late-stage bipolar disorder. Int J Neuropsychopharmacol. 2009 May;12(4):447-58. doi: 10.1017/S1461145708009310. Epub 2008 Sep 4. PMID 18771602
- [Background] Cheng LC, Pastrana E, Tavazoie M, Doetsch F. miR-124 regulates adult neurogenesis in the subventricular zone stem cell niche. Nat Neurosci. 2009 Apr;12(4):399-408. doi: 10.1038/nn.2294. Epub 2009 Mar 15. PMID 19287386
- [Background] Liu C, Teng ZQ, Santistevan NJ, Szulwach KE, Guo W, Jin P, Zhao X. Epigenetic regulation of miR-184 by MBD1 governs neural stem cell proliferation and differentiation. Cell Stem Cell. 2010 May 7;6(5):433-44. doi: 10.1016/j.stem.2010.02.017. PMID 20452318
- [Background] Li B, Jiang Y, Xu Y, Li Y, Li B. Identification of miRNA-7 as a regulator of brain-derived neurotrophic factor/alpha-synuclein axis in atrazine-induced Parkinson's disease by peripheral blood and brain microRNA profiling. Chemosphere. 2019 Oct;233:542-548. doi: 10.1016/j.chemosphere.2019.05.064. Epub 2019 May 23. PMID 31185338
- [Background] Gupta N, Jadhav S, Tan KL, Saw G, Mallilankaraman KB, Dheen ST. miR-142-3p Regulates BDNF Expression in Activated Rodent Microglia Through Its Target CAMK2A. Front Cell Neurosci. 2020 May 21;14:132. doi: 10.3389/fncel.2020.00132. eCollection 2020. PMID 32508597
- [Background] Lian N, Niu Q, Lei Y, Li X, Li Y, Song X. MiR-221 is involved in depression by regulating Wnt2/CREB/BDNF axis in hippocampal neurons. Cell Cycle. 2018;17(24):2745-2755. doi: 10.1080/15384101.2018.1556060. Epub 2018 Dec 27. PMID 30589396
- [Background] Lulli V, Buccarelli M, Ilari R, Castellani G, De Dominicis C, Di Giamberardino A, D Alessandris QG, Giannetti S, Martini M, Stumpo V, Boe A, De Luca G, Biffoni M, Marziali G, Pallini R, Ricci-Vitiani L. Mir-370-3p Impairs Glioblastoma Stem-Like Cell Malignancy Regulating a Complex Interplay between HMGA2/HIF1A and the Oncogenic Long Non-Coding RNA (lncRNA) NEAT1. Int J Mol Sci. 2020 May 20;21(10):3610. doi: 10.3390/ijms21103610. PMID 32443824
- [Background] Visitchanakun P, Tangtanatakul P, Trithiphen O, Soonthornchai W, Wongphoom J, Tachaboon S, Srisawat N, Leelahavanichkul A. Plasma miR-370-3P as a Biomarker of Sepsis-Associated Encephalopathy, the Transcriptomic Profiling Analysis of Microrna-Arrays From Mouse Brains. Shock. 2020 Sep;54(3):347-357. doi: 10.1097/SHK.0000000000001473. PMID 31743302
- [Background] Yuan H, Mischoulon D, Fava M, Otto MW. Circulating microRNAs as biomarkers for depression: Many candidates, few finalists. J Affect Disord. 2018 Jun;233:68-78. doi: 10.1016/j.jad.2017.06.058. Epub 2017 Jun 27. PMID 28673667
- [Background] Rubinsztein JS, Michael A, Paykel ES, Sahakian BJ. Cognitive impairment in remission in bipolar affective disorder. Psychol Med. 2000 Sep;30(5):1025-36. doi: 10.1017/s0033291799002664. PMID 12027040
- [Background] Martinez-Aran A, Vieta E, Colom F, Torrent C, Sanchez-Moreno J, Reinares M, Benabarre A, Goikolea JM, Brugue E, Daban C, Salamero M. Cognitive impairment in euthymic bipolar patients: implications for clinical and functional outcome. Bipolar Disord. 2004 Jun;6(3):224-32. doi: 10.1111/j.1399-5618.2004.00111.x. PMID 15117401
- [Background] Simonsen C, Sundet K, Vaskinn A, Birkenaes AB, Engh JA, Hansen CF, Jonsdottir H, Ringen PA, Opjordsmoen S, Friis S, Andreassen OA. Neurocognitive profiles in bipolar I and bipolar II disorder: differences in pattern and magnitude of dysfunction. Bipolar Disord. 2008 Mar;10(2):245-55. doi: 10.1111/j.1399-5618.2007.00492.x. PMID 18271903
- [Background] Summers M, Papadopoulou K, Bruno S, Cipolotti L, Ron MA. Bipolar I and bipolar II disorder: cognition and emotion processing. Psychol Med. 2006 Dec;36(12):1799-809. doi: 10.1017/S0033291706008804. Epub 2006 Aug 29. PMID 16938147
- [Background] Harkavy-Friedman JM, Keilp JG, Grunebaum MF, Sher L, Printz D, Burke AK, Mann JJ, Oquendo M. Are BPI and BPII suicide attempters distinct neuropsychologically? J Affect Disord. 2006 Aug;94(1-3):255-9. doi: 10.1016/j.jad.2006.04.010. Epub 2006 Jun 5. PMID 16750271
- [Background] Lee CY, Wang LJ, Lee Y, Hung CF, Huang YC, Lee MI, Lee SY. Differentiating bipolar disorders from unipolar depression by applying the Brief Assessment of Cognition in Affective Disorders. Psychol Med. 2018 Apr;48(6):929-938. doi: 10.1017/S003329171700229X. Epub 2017 Aug 22. PMID 28826415
- [Background] Lee SY, Wang LJ, Chang CH, Wu CC, Chen HL, Lin SH, Chu CL, Lu T, Lu RB. Serum DHEA-S concentration correlates with clinical symptoms and neurocognitive function in patients with bipolar II disorder: A case-controlled study. Prog Neuropsychopharmacol Biol Psychiatry. 2017 Mar 6;74:31-35. doi: 10.1016/j.pnpbp.2016.11.006. Epub 2016 Nov 30. PMID 27914864
- [Background] Pridmore S, Fernandes Filho JA, Nahas Z, Liberatos C, George MS. Motor threshold in transcranial magnetic stimulation: a comparison of a neurophysiological method and a visualization of movement method. J ECT. 1998 Mar;14(1):25-7. PMID 9661090
- [Background] Keefe RS, Fox KH, Davis VG, Kennel C, Walker TM, Burdick KE, Harvey PD. The Brief Assessment of Cognition In Affective Disorders (BAC-A):performance of patients with bipolar depression and healthy controls. J Affect Disord. 2014 Sep;166:86-92. doi: 10.1016/j.jad.2014.05.002. Epub 2014 May 11. PMID 25012414
- [Background] Lee CY, Lee SY, Huang YC, Hung CF, Lee Y, Lee MI, Wang LJ. The Chinese version of the Brief Assessment of Cognition in Affective Disorders: normative data of a Mandarin-speaking population. Clin Neuropsychol. 2018 Jan-Dec;32(sup1):1-14. doi: 10.1080/13854046.2017.1400108. Epub 2017 Nov 6. PMID 29108470
- [Background] Wang LJ, Lin PY, Lee Y, Huang YC, Hsu ST, Hung CF, Chen CK, Chen YC, Wang YL, Tsai MC. Validation of the Chinese version of Brief Assessment of Cognition in Schizophrenia. Neuropsychiatr Dis Treat. 2016 Oct 31;12:2819-2826. doi: 10.2147/NDT.S118110. eCollection 2016. PMID 27826194
- [Background] Li Z, Wang Z, Zhang C, Chen J, Su Y, Huang J, Yi Z, Yuan C, Hong W, Wang Y, Wu Z, Hu Y, Cao L, Peng D, Guan Y, Zou Y, Yu S, Cui D, Fang Y. Reduced ENA78 levels as novel biomarker for major depressive disorder and venlafaxine efficiency: Result from a prospective longitudinal study. Psychoneuroendocrinology. 2017 Jul;81:113-121. doi: 10.1016/j.psyneuen.2017.03.015. Epub 2017 Mar 18. PMID 28441588
- [Background] Zeger SL, Liang KY, Albert PS. Models for longitudinal data: a generalized estimating equation approach. Biometrics. 1988 Dec;44(4):1049-60. PMID 3233245